CLINICAL TRIAL: NCT00894062
Title: ComparisiOn of Neointimal coVerage betwEen zotaRolimus Eluting Stent and Everolimus Eluting Stent Using Optical Coherence Tomography at 9 Months (COVER OCT)
Brief Title: Comparison of Neointimal Coverage Between Zotarolimus Eluting Stent and Everolimus Eluting Stent
Acronym: COVER OCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Kim, Jung-Sun, MD, Ph D, Severance Hospital, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0483
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ZES resolute (Endeavor® resolute)
  Interventions: Device: Zotarolimus eluting stent (Endeavor resoulte - ZES resolute)
- 2 (Active Comparator): EES (Xience®)
  Interventions: Device: Everolimus eluting stent (Xience - EES)

INTERVENTIONS:
Device: Zotarolimus eluting stent (Endeavor resoulte - ZES resolute) — Zotarolimus eluting stent (ZES)
  Arms: 1
Device: Everolimus eluting stent (Xience - EES) — Everolimus eluting stent (EES)
  Arms: 2

SUMMARY:
Stent thrombosis is an important issue in drug eluting stents. Incomplete endothelial coverage and neointimal coverage over strut after drug eluting stent (DES) implantation could be a possible cause of stent thrombosis. Therefore, theoretically dual antiplatelet therapy should be continued to prevent the stent thrombosis until complete reendothelialization. But, detection of endothelial coverage over stent is not possible with the available intravascular devices in clinical practice. Among currently available intravascular devices, intravascular optical coherence tomography (OCT) could give a more clear identification for a thin layer of neointima with high-resolution (10-20 μm) compared to intravascular ultrasound (100-150 μm). Previous OCT studies showed the significant different pattern of neointimal coverage between bare metal stent (BMS) and DES. In the investigators' experience, there were also some differences in neointimal coverage among the DESs, especially zotarolimus eluting stent (ZES). ZES has been known to be associated with significantly more neointimal coverage than SES at 8 months intravascular ultrasound (IVUS). Both everolimus eluting stent (EES) and ZES resolute were recently introduced. The efficacy to suppress the neointimal growth for ZES resolute and EES might be improved, but safety for neointimal coverage needs to evaluate in human coronary artery. Therefore, this study will investigate the pattern of neointimal coverage over stent in ZES resolute and EES at 9 months after stent implantation.

DETAILED DESCRIPTION:
Recent autopsy study showed the most important histological and morphometric predictors of stent thrombosis were endothelial coverage and the ratio of uncovered to total strut after drug eluting stent (DES) implantation. Although there have been some controversies, incomplete stent apposition might be possible cause of very late stent thrombosis after DES implantation. Therefore, theoretically dual antiplatelet therapy should be continued to prevent the stent thrombosis until complete reendothelialization. But, detection of endothelial coverage over stent are no possible with available intravascular devices in clinical practice. Among currently available intravascular devices, intravascular optical coherence tomography (OCT) could give a more clear identification for a thin layer of NIH and malapposition with high-resolution (10 -20 μm) compared to intravascular ultrasound (100-150 μm). Previous OCT studies showed the significant different pattern of neointimal coverage between bare metal stent (BMS) and DES. In our experience, there was also some differences in neointimal coverage among the DESs, especially zotarolimus eluting stent (ZES). ZES have been known to be associated with significantly more neointimal coverage than SES at 8 months intravascular ultrasound (IVUS). This finding might be related with strut thickness and drug elution property. In our data, neointima was covered at 99.7% of stent strut in ZES, but 93.2% in sirolimus eluting stent (SES) at 9 month follow OCT. This difference was more distinct in patients with acute myocardial infarction (99.3% in ZES vs.79.9% in SES).

Both everolimus eluting stent (EES) was recently introduced and ZES resolute also will be available in the near future in Korea. Previous phosphorylcholine polymer was replaced with new, proprietary polymer which can provide extended elution kinetics in ZES resolute. Therefore, efficacy to suppress the neointimal growth might be improved but, safety for neointimal coverage needs to evaluate in human coronary artery. Both new DESs are cobalt chromium stent with thin stent strut and reported similar efficacy for suppressing the neointima growth. Also, endothelial coverage over stent strut occurred earlier compared to previous DESs (SES or PES) in animal experiments. But, there has been no data for neointimal coverage and malapposition of ZES resolute and EES using OCT in human coronary artery.

Recent paper according to Kubo et al reported that serial OCT examinations demonstrated markedly different vascular response up to 9 months after SES implantation between unstable angina and stable angina patients. These findings implied that initial native vessel status, which covered with stent, might be important and related with neointimal coverage and malapposition. But, there is little data evaluated the relationship between initial lesion status and neointimal coverage or late malapposition with OCT.

Therefore, this study investigates: 1) the relationship of the initial lesion and neointimal coverage or late malapposition and 2) the neointimal coverage and malapposition at 9 month after ZES resolute and EES implantation and 3) compare them between ZES resolute and EES at 9 months after stent implantation.

Study Objectives:

This study is a prospective open labeled randomized study to compare the neointimal coverage of ZES resolute (Endeavor® resolute) and EES (Xience®) in 9 month after stent implantation by OCT.

1. Primary end point:

   * The primary endpoint is to compare the neointimal coverage of ZES resolute (Endeavor® resolute) and EES (Xience®) at 9 months after stent implantation by OCT.
2. Secondary end points:

   * To investigate the relationship between initial lesion and neointimal coverage and malapposition at 9 months, and
   * To compare of neointimal growth between ZES resolute and EES at 9 months and to compare the difference in early and late malapposition between ZES resolute and EES at 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Significant coronary de novo lesion (> 70% by quantitative angiographic analysis)
* Patients with stable or acute coronary syndrome considered for coronary revascularization
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* The criteria for exclusion were contraindication to anti-platelet agents
* Proximal lesion within 15 mm from ostium
* Different DES in other vessel simultaneously
* Creatinine level 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy 1 year
* Complex lesion morphologies (aorto-ostial, bifurcation with > 2.0 mm side branch, unprotected left main, thrombus, severe calcification, chronic total occlusion)
* Target lesion is vein graft lesion
* Reference vessel < 2.5 mm or > 4.0 mm diameter by visual
* Long lesion that require more than two stents

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12

PRIMARY OUTCOMES:
Evaluation of neointimal coverage of ZES resolute (Endeavor® resolute) and EES Xience®) by OCT. | at 9 months after stent implantation

SECONDARY OUTCOMES:
Investigate the relationship between initial lesion and neointimal coverage and malapposition at 9 months. | 9 months after stent implantation
Comparison of neointimal growth between ZES resolute and EES at 9 months. | 9 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Kim, MD, Ph D, Principal Investigator — Division of Cardiology, Cardiovascular Hospital, Yonsei University
Locations (3):
- South Korea (3):
  - Dongsan Medical Center, Keimyung University, Daegu
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Kim JS, Kim BK, Jang IK, Shin DH, Ko YG, Choi D, Hong MK, Cho YK, Nam CW, Hur SH, Choi JH, Song YB, Hahn JY, Choi SH, Gwon HC, Jang Y. ComparisOn of neointimal coVerage betwEen zotaRolimus-eluting stent and everolimus-eluting stent using Optical Coherence Tomography (COVER OCT). Am Heart J. 2012 Apr;163(4):601-7. doi: 10.1016/j.ahj.2011.10.016. PMID 22520526